CLINICAL TRIAL: NCT03610061
Title: Phase I Dose Escalation Study of Radiotherapy and Durvalumab in Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL) and Follicular Lymphoma (FL): The RaDD Study
Brief Title: A Trial of Radiotherapy and Durvalumab in DLBCL and FL
Acronym: RaDD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: Olivia Newton-John Cancer Research Institute (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Eliza Hawkes, Chief Investigator, Austin Health
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2017-003-DV-008259; TRP16-006 (Other Grant/Funding Number: Victorian Cancer Agency)
Record Dates: First submitted 2017-11-14; First posted 2018-08-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Large B Cell Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy plus Durvalumab (Experimental): A minimum of 3 patients will initially be enrolled in each cohort of this arm. Patients will be allocated to a radiotherapy dose and site cohort from the schedule at registration. There will be no intra-patient dose or site escalations.
  Cohorts will escalate in number of anatomical sites of radiotherapy and dose of radiotherapy given subject to safety. Durvalumab will be administered at a fixed dose every 4 weeks IV.
  Interventions: Drug: Durvalumab; Radiation: Radiotherapy; Radiation: Radiotherapy (cohort 6 only)

INTERVENTIONS:
Drug: Durvalumab — All patients will receive:
  Day 1-Day 5: External Beam Radiotherapy to target site(s)-daily for 5 days (i.e. 5 fractions).
  D2: Commence durvalumab. Continue 4-weekly until disease progression. Patients can continue until a second radiological progression if clinical benefit is ongoing.
  Other Names: MEDI4736
Radiation: Radiotherapy — All patients will receive:
  Day 1-Day 5: External Beam Radiotherapy to target site(s)-daily for 5 days (i.e. 5 fractions).
  D2: Commence durvalumab. Continue 4-weekly until disease progression. Patients can continue until a second radiological progression if clinical benefit is ongoing.
Radiation: Radiotherapy (cohort 6 only) — Cohort 6 patients (only) will receive:
  Day 8-Day 10: External Beam Radiotherapy to target site(s)- daily (ie. 5 further fractions to a total of 10 fractions)

SUMMARY:
The primary objective for this study is to determine the safety profile of radiotherapy and durvalumab, a PD-L1 inhibitor.

Primary endpoint:

Toxicity, drug pharmacokinetics (PK), maximum tolerated dose (MTD) and recommended phase two dose (RPTD) of simultaneous radiotherapy plus durvalumab in patients with relapsed or refractory DLBCL or FL.

Secondary endpoints:

* ORR
* Progression-free survival
* Overall survival

Exploratory endpoints include description of biological effects of combination radiotherapy plus durvalumab (Imaging results, immune function, PK and PD-see 'research methodologies') and in the PET-Sub-Study, biodistribution of 89Zr Durvalumab and 89Zr-IAB22M2C.

DETAILED DESCRIPTION:
Diffuse large B cell lymphoma (DLBCL) and Follicular Lymphoma (FL) are the most common non Hodgkin lymphomas. Standard first line treatment achieves cure in approximately half of patients. However 30% die from relapsed lymphoma.

Durvalumab (an antibody which blocks programmed cell death ligand 1) and other immunotherapies fight cancer by blocking barriers to immune system activity. Immune control of lymphoma provides the prospect of cure, even when chemotherapy has failed. Radiotherapy has striking effects on the immune system and can boost responses to these immunotherapies. The effect of concurrent radiotherapy and durvalumab in DLBCL and FL is unproven.

This study will evaluate the safety and effect of simultaneous radiotherapy plus durvalumab (a PD-L1 inhibitor) in relapsed DLBCL and FL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects aged 18 years weighing more than 30 kg
2. Histologically proven CD20-positive relapsed or refractory diffuse large B cell non-Hodgkin lymphoma (DLBCL) either de novo or DLBCL transformed from any indolent B-non-Hodgkin lymphoma (including Richter's transformation) Or follicular lymphoma grade 1-3A, or Grade 3B, according to the current World Health Organization classification on tissue biopsy. Archived tissue is permitted however must have been obtained after the last known therapy. The Trial Management Group retains the option to limit the number of participants enrolled with a specific histology.
3. At least 1 line of previous treatment for lymphoma which must include a CD20 monoclonal antibody such as rituximab, with no curative option as determined by the investigator. Prior radiotherapy is permitted.
4. Patients with DLBCL must not be eligible or willing to receive high-dose (myeloablative) chemotherapy (HDC) and autologous stem cell transplant (ASCT) OR has received prior ASCT.
5. Eastern Collaborative Oncology Group performance status 0, or 1, unless attributable to lymphoma in which case patients of performance status 2 are also eligible.
6. Patients must have measurable disease (at least one bi-dimensionally measurable site of disease that has not been previously irradiated OR has progressed after radiotherapy: nodal disease >1.5 cm or an extranodal lesion > 1.0 cm in longest perpendicular diameter). At least three disease sites must be FDG-avid on PET imaging AND amenable to radiotherapy according to local radiation oncology investigator review.
7. One site of disease must be amenable to biopsy. It is preferable that this is a site not planned for radiotherapy, but not mandated. A fresh tumor biopsy collected during screening and /or archival tumor tissue collected after the last relapse/disease progression (material which has been collected before the last line of treatment is not accepted). In addition, a sufficient amount of the material is required for acceptance of the archival material. If neither condition occurs, a fresh tumor biopsy needs to be performed as stated above.
8. Adequate bone marrow function with platelets > 50 x109/l; neutrophils > 1.0x109/l at the time of study entry unless attributed to bone marrow infiltration by lymphoma.
9. Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method).
10. Adequate hepatic function defined by a total bilirubin level ≤ 2 × the upper limit of normal (ULN) range (excluding Gilbert's disease where a level of ≤ 3 ×ULN is acceptable) and AST and alanine aminotransferase (ALT) levels ≤ 2.5 × upper limit of institutional normal range unless attributed to lymphoma.
11. No concurrent uncontrolled medical condition as determined by the investigator.
12. Life expectancy > 3 months.
13. Negative blood pregnancy test at screening for women of childbearing potential. Effective contraception for both male and female subjects if the risk of conception exists.

(Note: The effects of the trial drug on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use effective contraception, defined as 2 barrier methods, or 1 barrier method with an intrauterine device, or use of oral female contraceptive. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately. Effective contraception at least 30 days prior and up to 3 months after treatment is required for all women of childbearing potential and male subjects will be advised not to father a child during the 3 months after treatment completion. Male subjects will be requested to seek advice on conservation of sperm prior to treatment.) n) Signed written informed consent before any trial-related procedure is undertaken that is not part of the standard patient management.

Exclusion Criteria:

1. T-cell lymphoma, Hodgkin lymphoma.
2. Central nervous system, meningeal or spinal cord involvement by lymphoma.
3. Prior therapy with any antibody or drug targeting T-cell coregulatory proteins (immune checkpoints) such as PD-1, PD-L1, or cytotoxic T-lymphocyte antigen-4 (CTLA-4).
4. Patients with active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

i) Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible ii) Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day iii) Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable.

e) Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion: i. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) ii. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisolone or its equivalent iii. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

.iv.Patients requiring steroids for symptom control during the screening period may receive a single course of prednisolone at a dose of up to 100mg daily (or equivalent) for a maximum of 5 days at the discretion of the local PI. Steroids must not be given within 5 days of radiotherapy. Note that steroids are optimally avoided due to the potential for reduction in durvalumab activity

f) Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma) g) Past history of interstitial lung disease. h) Prior organ transplantation, including allogeneic stem-cell transplantation i) Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

j) Major surgery for any reason, except diagnostic biopsy, within 4 weeks of enrolment and/or if the subject has not fully recovered from the surgery within 4 weeks of enrolment k) Any other serious active disease, including but not limited to; i) clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina pectoris, congestive heart failure (New York Heart Association Classification Class ≥ II), or serious cardiac arrhythmia requiring medication (including QTc prolongation of > 470 ms and/or pacemaker) or prior diagnosis of congenital long QT syndrome.

ii) uncontrolled active infection, iii) uncontrolled diabetes (e.g., haemoglobin A1c ≥ 8.5%) l) Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive) m) Medical or psychiatric conditions that compromise the patient's ability to give informed consent.

o) Subject is pregnant, lactating or unwilling/unable to use adequate contraception p) Subject weighs less than 30kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Number of participants treated with radiotherapy and durvalumab with treatment-related adverse events as assessed using CTCAE v4.0. To determine the maximum tolerated dose (MTD). | First 28 days of treatment
  A minimum of 3 patients will initially be enrolled in each cohort, if none of the first 3 patients experiences a dose limiting toxicity (DLT), the doses in that cohort will be deemed safe and tolerable and escalation may continue. DLTs will be grade 4 neutropenia or thrombocytopenia, grade 3 hemolysis, grade 4 immune related AEs.
  If 1 of the first 3 evaluable patients in a cohort experiences a DLT, the cohort will be expanded to at least 6 patients. If there are no further DLTs in the first 6 DLT-evaluable patients, the doses in that cohort will be deemed safe and tolerable and escalation may continue.
  If a DLT is observed in ≥ 33% of patients (e.g., 2 or more of up to 6 patients), the dose combination at which this occurs will be considered intolerable and the MTD will have been exceeded for radiotherapy If the MTD is exceeded in any cohort, the highest dose combination at which fewer than 33% experience a DLT will be declared the combination MTD.

SECONDARY OUTCOMES:
Response rates (according to the Lugano classification for Response Criteria for Non-Hodgkin Lymphoma) | 0-12 months
  Response rates
Progression free survival | From ceasing treatment annually up to 5 years
  Progression free survival in patients who cease treatment due to toxicity.
Overall survival | Every 6 months from PD up to two years.
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Hawkes, MD, Principal Investigator — Austin Health
Locations (3):
- Australia (3):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
IPD is the property of the Sponsor (Olivia Newton John Cancer Research Institute). Results from the research intends to be published/presented in relevant publications/conferences for colleague review

REFERENCES:
- [Derived] Hawkes EA, Palmer JB, Khor R, Lee ST, Burgess M, Law SC, Gandhi MK, Chong G, Shortt J, Chowdhury R, Swain F, Churilov L, MacManus M, Smith C, Scott FE, Martynchyk A, Barraclough A, Manos K, Scott AM, Keane C. T-cell dysregulation informs radiotherapy-immunotherapy response in B-cell lymphoma: results from a phase 1 trial. Blood Adv. 2025 Oct 28;9(20):5263-5273. doi: 10.1182/bloodadvances.2025016505. PMID 40540795